CLINICAL TRIAL: NCT04413435
Title: Clinical Characteristics of Critically Ill Patients With 2019 Novel Coronavirus (COVID-19): Do We Need a New Triage System?
Brief Title: Clinical Characteristics of Critically Ill Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Nevsehir Public Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif Yazar, Specialist, Nevsehir Public Hospital
Other Study IDs: 2020-245
Record Dates: First submitted 2020-05-25; First posted 2020-06-04 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Coronavirus Infection; Critical Illness; Characteristics Disease
MeSH Terms: conditions — Coronavirus Infections; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Confirmed COVID-19 cases: Patients with PCR test positive were considered as the confirmed COVID-19 cases.
  Interventions: Other: File Scanning
- Suspected COVID-19 cases: The suspected COVID-19 cases were defined as follows: those who were interpreted in favor of the suspected covid-19 on c-CT by radiologists in addition to the typical symptoms of the novel coronavirus disease such as cough, high fever (>38,5 °C), or dyspnea, and those with a history of contact with another confirmed COVID-19 patient in addition to typical symptoms.
  Interventions: Other: File Scanning

INTERVENTIONS:
Other: File Scanning — The patients' epidemiological, clinical, laboratory, and radiological characteristics and treatment and outcomes data will accessed from Hospital Data Management System (HDMS) of Konya Training and Research Hospital and Public Health Management System (PHMS) of Ministry of Health.

SUMMARY:
Critically ill patients with COVID-19 have hospitalized in an ICU due to the closer monitoring and therapy. In fact, ICU admissions are dependent on the severity of illness and the ICU capacity of the health-care system. Hence, it may be need a new scoring system for contagious critically ill patients.

DETAILED DESCRIPTION:
Critically ill patients with COVID-19 have hospitalized in an ICU due to the closer monitoring and therapy. In fact, ICU admissions are dependent on the severity of illness and the ICU capacity of the health-care system. Therefore, many patients with confirmed COVID-19 with RT-PCR and/or suspected COVID-19 were hospitalized in ICUs with a limited number of beds. This ambiguity can result in both contamination risk to uninfected patients and occupancy rate of the limited ICU beds. Hence, it may be need a new scoring system for contagious critically ill patients. The aim of this study was to describe the epidemiological and clinical features of 75 critically ill patients due to COVID-19 and to compare confirmed COVID-19 cases with suspected COVID-19 cases in our critical care units.

ELIGIBILITY:
Inclusion Criteria:

* All patients with confirmed COVID-19 and suspected COVID-19

Exclusion Criteria:

* All patients <18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — patients >18 years old
Study Population: All patients with confirmed COVID-19 and suspected COVID-19 patients who hospitalized in ICUs allocated for patients with novel coronavirus disease.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Polymerase Chain Reaction (PCR) test | 5 days
  To compare confirmed COVID-19 cases with suspected COVID-19 cases in critical care units.

SECONDARY OUTCOMES:
A scoring system for patients to be admitted to the intensive care unit | 5 days
  To use symptoms, medical history, computed tomography and laboratory examinations for scoring system to detect suspected COVID-19 cases admitted to the intensive care units.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Trainig and Research Hospital, Konya, Turkey (Türkiye)